CLINICAL TRIAL: NCT04301778
Title: A Phase II Study of Durvalumab (MEDI4736) in Combination With a CSF-1R Inhibitor (SNDX-6532) Following Chemo or Radio-Embolization for Patients With Intrahepatic Cholangiocarcinoma.
Brief Title: Durvalumab and SNDX-6532 Following Chemo or Radio-Embolization for Patients With Intrahepatic Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Syndax Pharmaceuticals (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2031; IRB00233351 (Other: Johns Hopkins Institutional Review Board)
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Results first posted 2023-03-31 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Unresectable Intrahepatic Cholangiocarcinoma
Keywords: colony stimulating factor -1 receptor (CSF-1R) inhibitor; Anti-PD-1 (receptor blocking antibody); Immunotherapy; Intra-arterial therapy; Y90 (yttrium-90 radioembolization); conventional transarterial chemoembolization (cTACE); Chemo-embolization; Radio-embolization; Biliary tract; Intrahepatic Cholangiocarcinoma; Monoclonal antibody
MeSH Terms: conditions — Cholangiocarcinoma | interventions — durvalumab; axatilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab and SNDX-6352 (Experimental): Participants will receive Durvalumab and SNDX-6352.
  Interventions: Drug: Durvalumab; Drug: SNDX-6352

INTERVENTIONS:
Drug: Durvalumab — 1. Durvalumab - 1500 mg via IV infusion over 60 minutes (-5/+10 min) on day 1 of each 28-day cycle (every 4 weeks).
  2. Drug - 1500mg IV
  Other Names: MEDI4736
Drug: SNDX-6352 — 1. SNDX-6352 - 3mg/kg via IV infusion over 30 minutes (-5/+10 min) on days 1 and 15 of each 28-day cycle (every 2 weeks), starting with cycle 2 (not given during cycle 1).
  2. Drug - 3mg/kg IV
  Other Names: UCB6352

SUMMARY:
The purposed of this research is to study the safety and clinical activity of the combination of durvalumab and a CSF-1R inhibitor (SNDX-6352) in people with Intrahepatic Cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Have cytologically confirmed intrahepatic cholangiocarcinoma.
* All disease must be localized to the liver (locally advanced).
* Subjects must not be deemed surgical candidates.
* Must be a candidate for conventional transarterial chemoembolization or yttrium-90 radioembolization.
* Must have measureable disease be mRECIST. Measurable disease will be confirmed by radiological imaging (MRI, CT).
* Age ≥18 years
* Body weight > 30 kg
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Life expectancy ≥12 weeks.
* Patient must have adequate organ function defined by the study-specified laboratory tests as per the protocol.
* Child Pugh Class A
* Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine clearance CL>40 mL/min by the Cockcroft-Gault formula.
* Woman of childbearing potential must have a negative pregnancy test and follow contraceptive guidelines as defined per protocol.
* Must use acceptable form of birth control while on study.
* Men must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.
* Willing and able to comply with the protocol for the duration of the study

Exclusion Criteria:

* Candidate for surgical resection
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up of an interventional study.
* Major surgery within 4 weeks prior to initiation of study treatment.
* Received the last dose of anticancer therapy ≤ 28 days prior to the first dose of study drug.
* All toxicities NCI CTCAE Grade ≥2 attributed to prior anti-cancer therapy other than alopecia, vitiligo, and neuropathy.
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment.
* History of allogenic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, checkpoint inhibitor-induced immune mediated reaction or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]).
* Patient with uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant muscle disorders or psychiatric illness/social situations that would limit compliance with study requirements.
* History of known additional primary malignancies.
* History of leptomeningeal carcinomatosis.
* Brain metastases or spinal cord compression.
* History of active primary immunodeficiency.
* Infection with Tuberculosis, HIV or hepatitis B or C at screening.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of treatment.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.
* Pregnant or breastfeeding women.
* Has a history of allergy to study treatments or any of its components of the study.
* Prior randomization or treatment in a previous durvalumab and/or SNDX-6532 clinical study regardless of treatment arm assignment.
* Patient has clinically significant heart disease.
* Any other sound medical, psychiatric, and/or social reason as determined by the Investigator.
* Unwilling or unable to follow the study schedule for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2024-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zheng, MD, Principal Investigator — Sidney Kimmel Cancer Center at the Johns Hopkins Medical Institution
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Durvalumab and SNDX-6352: Participants received Durvalumab and SNDX-6352.
  Durvalumab: 1500 mg IV over 60 minutes on day 1 of each 28-day cycle (every 4 weeks).
  SNDX-6352: 3mg/kg IV over 30 minutes on days 1 and 15 of each 28-day cycle (every 2 weeks), starting with cycle 2 (not given during cycle 1).
Period: Overall Study
Arm/Group | Durvalumab and SNDX-6352
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Durvalumab and SNDX-6352
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 60 [39 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG scale measures performance status, with scores ranging from 0-5; 0= fully active, performs without restriction, 1= can ambulate, but restricted in physically strenuous activity, 2= ambulatory and capable of self-care, but unable to work, active for >50% of waking hours, 3= limited self-care, confined to bed or chair for >50% of waking hours, 4= completely disabled, totally confined to bed/chair, 5= deceased
  Participants
    ECOG 0 | 4
    ECOG 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per mRECIST (Modified RECIST)
Description: ORR is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on the Response Evaluation Criteria in Solid Tumors (mRECIST) at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab and SNDX-6352
Number analyzed (Participants) | 5
Participants | 1

2. Primary Outcome: Number of Participants Experiencing Study Drug-related Toxicities
Description: Number of participants who experience treatment related adverse events ≥ grade 3 as defined by CTCAE 5.0.
Time Frame: up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab and SNDX-6352
Number analyzed (Participants) | 5
Participants | 2

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the number of months from the start of study treatment to time of death. Individuals are censored at the date of the last contact if no event occurs. The estimation method used was Kaplan-Meier.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab and SNDX-6352
Number analyzed (Participants) | 5
months | 15.3 [14.2 to NA] — upper limit not reached

4. Secondary Outcome: Progression-free Survival (PFS) Per mRECIST
Description: PFS is defined as the number of months from the date of treatment to disease recurrence [disease recurrence (DR) progressive disease (PD) or relapse from complete response (CR) as assessed using mRECIST criteria] or death due to any cause. Per mRECIST criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Time Frame: 8 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab and SNDX-6352
Number analyzed (Participants) | 5
months | 3.6 [1.8 to NA] — upper limit not reached

5. Secondary Outcome: Duration of Response (DOR)
Description: Number of days from the start of partial response (PR) or complete response (CR) by radiographic scans, whichever is recorded first, until the first date that progressive disease or death is documented. Per mRECIST, CR = disappearance of any intratumoral arterial enhancement in all target lesions, PR is =>30% decrease in sum of diameters of target lesions.
Time Frame: 8 months
Population: Only patients with either a partial or complete response by mRECIST are included in the analysis.
Measure: Number; unit: days
Arm/Group | Durvalumab and SNDX-6352
Number analyzed (Participants) | 1
days | 57

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of study drug until 90 days from last dose of study drug, up to 1 year. Patients were followed for survival (all-cause mortality) for up to 2 years
Description: Adverse reporting collection was conducted by regular investigator assessment and laboratory measurements.
Arm/Group | Durvalumab and SNDX-6352
All-Cause Mortality (participants affected / at risk) | 4/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab and SNDX-6352 (N=5)
Skin infection (Infections and infestations) | 1 (1)
Ruptured femoral pseudoaneurysm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab and SNDX-6352 (N=5)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (6)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (2)
Edema limbs (General disorders) | 1 (1)
Generalized edema (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (5)
Pain at biopsy site (General disorders) | 2 (2)
ALT increased (Investigations) | 1 (1)
AST increased (Investigations) | 4 (8)
Blood LDH increased (Investigations) | 2 (3)
CPK increased (Investigations) | 4 (13)
Weight loss (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT04301778/Prot_SAP_000.pdf